CLINICAL TRIAL: NCT02418182
Title: A Randomized Controlled Trial of Oral Acetaminophen for Analgesic Control After Transvaginal Oocyte Retrieval
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Deidre D Gunn, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: F141003005
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pain
Keywords: Analgesic; Pain Control; IVF; Tylenol; Acetaminophen; Egg Retrieval; iv vitro Fertilization
MeSH Terms: conditions — Pain; Agnosia | interventions — Acetaminophen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Control group participants will receive unlabelled 2 non-active placebo tablets approximately 1 hour prior to transvaginal oocyte retrieval procedure.
  Interventions: Drug: placebo
- Experimental (Experimental): Experimental group participants will receive 2 acetaminophen 500mg tablets approximately 1 hour prior to transvaginal oocyte retrieval procedure.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen total dose of 1000mg
  Other Names: Tylenol; paracetamol
  Arms: Experimental
Drug: placebo — subjects randomized to this group will be given placebo tablets
  Other Names: sugar pill
  Arms: Control

SUMMARY:
Current standard of care is no pretreatment medications before the egg retrieval, and the investigators would like to evaluate if preoperative Tylenol improves procedure and post procedure pain control over the current practice (no pre-treatment). Specifically, this study will compare Tylenol with a placebo when given before retrieval procedures. The investigators believe that if Tylenol can offer better analgesic relief than no pretreatment medications, then it may reduce the amount of narcotics needed by patients during and after the procedure and contribute to better patient satisfaction. . This study will enroll 100 participants all from University of Alabama at Birmingham (UAB).

DETAILED DESCRIPTION:
The current standard of care for oocyte retrieval in IVF involves fentanyl, propofol, as well as oxycodone. However, there exists little data of alternatives to narcotic medications for analgesic purposes in oocyte retrieval procedures. A retrospective study published in 2013 showed potential for NSAID's, specifically ketorolac, to significantly improve pain scores in women undergoing oocyte retrieval. It was also shown that the use of these medications did not significantly alter pregnancy rate, live birth rate, or miscarriage rate in these patients. Few other studies have delved into the question of anesthetics for oocyte retrievals except a prospective study in 2006. This study shows that no significant difference in pregnancy rates of implantation occurs with the use of acetaminophen and diclofenac vs. acetaminophen alone if given post-operatively. However, pain was not measured in this study for either group. Therefore, it is clear that there exists limited data on the subject of analgesics used in oocyte retrievals for in vitro fertilization and that more exploration into alternative medications is required to find the most effective and least harmful option.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Undergoing Transvaginal Oocyte Retrieval Procedure

Exclusion Criteria:

* Acetaminophen allergy
* Opioid dependency

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deidre D Gunn, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Deidre D Gunn, MD, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan
Supporting Information: Study Protocol, SAP
Time Frame: To Be Determined
Access Criteria: Shared through CT.gov

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Experimental
Started | 49 | 50
Completed | 31 | 33
Not Completed | 18 | 17
Not completed — Unable to re-consent | 18 | 15
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Of 99 patients enrolled, 72 required re-consent. Of these, 39 re-consented and 33 could not be re-consented. Therefore, these 33 were excluded, leaving 66 patients for analysis. Two of these were lost to follow-up and were excluded, leaving 64 women (31 control, 33 active arm) in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (4.4) | 32 (5.0) | 32.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Median of Cumulative Pain Scores Up to 60 Minutes Post Procedure
Description: Median of cumulative pain scores (measured on a visual analog scale from 0-10 where 0=no pain and 10=worst pain) taken during the recovery period (15, 30, 45, and 60 minutes post procedure)
Time Frame: 60 minutes post-procedure
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 31 | 33
score on a scale | 2 [0 to 3] | 2 [1 to 4]

2. Primary Outcome: Median of Cumulative Pain Scores Up to 24 Hours Post Procedure
Description: Median Pain score (measured on a visual analog scale from 0-10 where 0=no pain and 10=worst pain) taken at 24-hours post-procedure
Time Frame: 24-hours post-procedure
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 31 | 33
score on a scale | 1 [0 to 2] | 2 [0 to 3]

3. Secondary Outcome: Number of Participants With Use of Analgesics up to 60 Minutes Post Procedure
Description: Number of participants requiring use of analgesic medications in the post-operative recovery suite
Time Frame: 60-minutes post-procedure
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 31 | 33
Participants | 11 | 18

4. Secondary Outcome: Number of Participants With Use of Analgesics in the First 24 Hours After Discharge
Description: Number of participants with use of analgesic medications in the first 24 hours after discharge from procedure
Time Frame: 60-minutes post-procedure to 24-hours after procedure
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 31 | 33
Participants | 25 | 27

ADVERSE EVENTS:
Time Frame: Each participant was measured from baseline through 24 hours post-procedure.
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 4/31 | 9/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=31) | Experimental (N=33)
Nausea/Vomiting (Gastrointestinal disorders) | 4 (4) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02418182/Prot_SAP_000.pdf